CLINICAL TRIAL: NCT01550107
Title: A Prospective Study to Evaluate the Effect of Allopurinol on Muscle Energetics in Primary Sarcopenia
Brief Title: Allopurinol in Functional Impairment (ALFIE) Trial: 'Improving Muscle Strength'
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Dr. Jacob George, Chief Investigator, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GEO006
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Allopurinol; Xanthine Oxidase; MR Spectroscopy
MeSH Terms: conditions — Sarcopenia | interventions — Allopurinol; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Active Comparator): Allopurinol 600mg tablets
  Interventions: Drug: Allopurinol
- Lactose tablets (Placebo Comparator): Placebo Lactose tablets
  Interventions: Drug: Lactose tablets

INTERVENTIONS:
Drug: Allopurinol — 300mg b.d for 24 weeks
  Arms: Allopurinol
Drug: Lactose tablets — matched placebo tablets b.d
  Arms: Lactose tablets

SUMMARY:
Sarcopenia is defined as the presence of low muscle mass and either decreased muscle strength or function. It is increasingly becoming a significant cause of frailty, loss of independence and physical disability in ageing western populations. Recent experimental evidence has revealed that skeletal muscle is particularly susceptible to damaging molecules that result in oxidative stress and that oxidative stress plays a prominent role in the development and progression of sarcopenia. The investigators have previously shown that the xanthine oxidase inhibitor allopurinol is able to abolish vascular oxidative stress and improve endothelial function in cohorts such as optimally treated chronic heart failure and chronic kidney disease. Recently, the investigators have also shown that allopurinol improves exercise tolerance and time to ST-depression in optimally treated coronary artery disease, suggesting that allopurinol could also exert its effects through ATP and/or oxygen sparing mechanisms.

Therefore, we propose a randomised double blind placebo-controlled parallel group trial of allopurinol in patients with primary sarcopenia using MR-spectroscopy and Flow Mediated Dilatation to investigate the possible mechanisms that underlie this exciting possibility

DETAILED DESCRIPTION:
this section will be completed once the study is officially recruiting

ELIGIBILITY:
Inclusion Criteria:

Age 65 and over 6-Minute Walk Distance <400m

Exclusion Criteria:

Documented history of peripheral arterial disease. Pre-existing diagnosis of severe heart failure (LVEF<35%). Malignancy under active treatment (excluding basal cell carcinoma). Severe COPD (Physician diagnosis). Intolerance to allopurinol. Individuals with Active Acute Gout currently taking allopurinol; or those who have stopped taking allopurinol ≤1month previously for this condition.

On long term high dose steroids (eq. Prednisolone>10mg/day due to risk of steroid induced myopathy and osteoporosis).

Immobility that would render the patient incapable of doing the Short Physical Performance Battery Test (SPPB) or 6MWT.

Patients who have participated in any other clinical drug trial within the previous 30 days will be excluded.

Cognitive impairment precluding informed consent. Any other considered by a study physician to be inappropriate for inclusion.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Improvement in Muscle energetics as measured by MR-spectroscopy | 24 weeks
  PCr repletion,Post-exercise muscle perfusion via arterial spin labelling (ASL) Pi/PCr ratio (a measure of ADP levels) Change in muscle volume (as measured by cross-sectional area on MR obtained during perfusion mapping)

SECONDARY OUTCOMES:
Short Performance Battery test | 24 weeks
6-Minute Walk Test | 24 weeks
Change in Flow Mediated Dilatation | 24 weeks
Markers of oxidative stress (F2-Isoprostanes) | 24 weeks
Quality of Life measured by EuroQOL EQ5D questionnaire | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacob George, MRCP MD, Principal Investigator — University of Dundee; Allan Struthers, MD FRCP, Study Director — University of Dundee; Marion McMurdo, MD FRCP, Study Director — University of Dundee; Miles Witham, PhD FRCP, Study Director — University of Dundee; Graeme Houston, FRCP FRCR, Study Director — University of Dundee; Steve Gandy, PhD, Study Director — University of Dundee; Peter Donnan, PhD FRSS, Study Director — University of Dundee; Clare Clarke, PhD MCSP, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee Medical School, Dundee, Angus, United Kingdom